CLINICAL TRIAL: NCT05092932
Title: Normative Research of Walking Aid Selection in Normal Subjects
Brief Title: Walking Aid Assessment, Arm Strength and Force Under the Foot in Normal Subjects
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Audrey Zucker-Levin, Professor, University of Saskatchewan
Other Study IDs: NER32
Record Dates: First submitted 2020-02-23; First posted 2021-10-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Physical Examination; Middle Age; Aged; Young Adult; Adolescent; Gait
Keywords: healthy; gait; plantar force; balance; muscle function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal Control Data: Normal adults with no history of neuromusculoskeletal disease will be recruited for this study. Participants will be independent walkers (no walking aid needed) and will not have needed a walking aid for injury over the past 5 years.
  Participants will walk 200 m under 4 randomized conditions: non-weightbearing ambulation using crutches, a walker, a wheeled knee walker, and unaided walking. An in-shoe sensor will measure stance limb plantar force, a stopwatch will time each walk, perceived exertion will be reported using the BORG CR-10 scale, and device preference will be identified.
  Interventions: Other: Normal Foot Force

INTERVENTIONS:
Other: Normal Foot Force — LoadSol Insoles will be inserted into the participants shoes. The device measures the pressure distribution on the bottom of the foot. Participants will then be asked to walk normally, use crutches, use a walker, and use a wheeled knee scooter. The pressure placed throughout the foot will be analyzed and compared under different conditions. This testing will take approximately 10 minutes.
  Other Names: Loadsol

SUMMARY:
This study will collect biomedical performance data on walking characteristics in normal, healthy people when walking with walking aids and when walking unaided. Data will be used for independent reporting and for comparison to matched people with pathological conditions. Data collected will including walking ability, balance, force under the feet when walking and muscle strength.

DETAILED DESCRIPTION:
Young adults often tolerate the increased energy expenditure, coordination, and stance limb discomfort associated with walking aids for non-weightbearing ambulation. It is not clear how walking aid selection affects stance limb plantar force, walking speed, perceived exertion, and device preference in adults over 50 years of age..

This project is a prospective randomized crossover study using healthy adults, aged over 50 years, with no use of walking aids within 5 years. Participants will walk 200 m under 4 randomized conditions: single non-weightbearing ambulation using crutches, a walker, a wheeled knee walker, and unaided walking. An in-shoe sensor will measure stance limb plantar force, a stopwatch will be used to time each walk, a hand held dynamometer will measure arm muscle strength, perceived exertion will be reported using the BORG CR-10 scale, and device preference will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Able bodied individuals self reported good health

Exclusion Criteria:

* recent fractures history of neurologic disease or events.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 200 healthy adults who independently walk with or without an assistive device.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Force under the stance limb foot | Through study completion, an average of one day. This is a one time assessment comparing differences in the normal force under the foot when the participant walks under 4 walking conditions.
  A wireless insole force sensor (LoadSol; Novel Inc) will be fitted in the shoe of the stance foot to measure stance limb plantar force during each walking trial. This force sensor covers the entire plantar surface of the foot and manufacturer's protocol for calibration will be applied for each participant before data is recorded at 100 Hz via Bluetooth connection to an iOS device (ie, an iPad).

SECONDARY OUTCOMES:
Arm strength in newtons | Through study completion an average of one day. This is a one time assessment to correlate strength with force under the stance limb foot with upper extremity strength under the 4 walking conditions.
  a hand held dynamometer will measure strength of the triceps, biceps, and latissimus Dorsi
Perceived Exertion | Through study completion, an average of one day. This is a one time assessment to compare perceived exertion when the participant walks under 4 walking conditions.
  The BORG revised category-ratio scale. Participants will be asked to rate the exertion from 0 "nothing at all" to 10 "maximal" after walking with each walking aid.
Walking aid preference | Through study completion, an average of one day.
  This is a one time assessment to determine which walking device is preferred after walking with all four devices.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey R Zucker-Levin, PhD, Principal Investigator — The University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada